## INFORMED CONSENT FORM

| I do hereby consent to the procedure being performed upon : |
|---|
| My Name : |
| CR Number : |
| The nature and extent of such a procedure, I have entirely to the discretion of Medical Officer performing the procedure. I have been informed about the risks of this procedure. I will not hold any of the hospital staff responsible for any risks involved in or accidents occurring during it or after the procedure. I do hereby voluntarily give consent for participation in this research project. |
| Date: |
| Patient's sign: |
| Patient's address: |
| Patient's CNIC: |
| Project Incharge: |

NO F.2-81/2020-GENL/ 428 7 Z
JINNAH POSTGRADUATE MEDICAL CENTRE
KARACHI.75510.

Dated the 7/52020

Dr. Faiza Shabbir Department of Dermatology W-10 JPMC, Karachi.

Subject:

A Randomized controlled trial of comparative efficacy of topical tazarotene Gel 0.1% versus microneedling in atrophic post-acne scars.

With reference to your application / letter dated 12<sup>th</sup> February, 2020, on the subject noted above and to say that the Institutional Review Board has approved your subject proposal.

Prof. A.R. Jamali Head of Department Orthopaedic Surgery and Chairman Institutional Review Board Committee JPMC, Karachi.

Copy forwarded for information and necessary action to:

Dr. Rabia Ghfoor, Assistant Prof. of Dermatology W-10, JPMC, Karachi.